CLINICAL TRIAL: NCT01329497
Title: The Effect of Systemic Dietary Instruction on Management of Plasma Phosphorus Levels in Peritoneal Dialysis (PD) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Huili Dai, Shanghai Jiaotong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: phosphorus
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2010-11

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- interventional group (Experimental)
  Interventions: Other: systemic dietary instruction

INTERVENTIONS:
Other: systemic dietary instruction — systemic dietary instruction based on continuous quality improvement (CQI) team-oriented approach

SUMMARY:
Hyperphosphatemia is highly prevalent in PD patients, and it is an independent risk factor for all-cause and cardiovascular mortality in these patients. Effective treatments are limited in suppressing plasma phosphorous. Because of the nearly linear relationship between protein and phosphorus intake, high dietary protein intake (DPI, 1.2-1.3g/kg/d recommended by KDOQI) would load high phosphorus burden in PD patients. It is suggested that hyperphosphatemia is hard to avoid under such a DPI level, even as the patients take sufficient phosphorus blinders and receive high PD dosage. The present study is to investigate whether systemic dietary instruction would show effects on control of hyperphosphatemia in PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Stable on PD for at least three month
2. Aged from 18 to 75 years old
3. Informed consent approval

Exclusion Criteria:

1. Malnutrition (based on SGA results)
2. Infection or inflammation within 1 month
3. Concurrent wasting disease (i.e. cancer, tuberculosis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Plasma phosphorus levels | up to 1 year

SECONDARY OUTCOMES:
Plasma calcium levels | up to one year
Carotid artery intima-media thicknesses | up to 1 year
Plasma albumin levels | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqi Qian, MD, Study Director — RenJi Hospital
Locations (1):
- Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China